CLINICAL TRIAL: NCT00270036
Title: A Double-Blind, Placebo-Controlled Study to Determine the Safety of r-HuEPO and Whether r-HuEPO Can Reduce Post-Operative Transfusion Requirements in Subjects Undergoing Major Orthopedic Surgery
Brief Title: A Study to Determine the Safety of Epoetin Alfa and Whether Epoetin Alfa Can Reduce the Need for Blood Transfusions in Patients After Major Orthopedic Surgery.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005902
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-11

CONDITIONS: Blood Transfusion; Orthopedic Procedures; Anemia
Keywords: Blood transfusion; epoetin alfa; epogen; erythropoietin; orthopedic procedures; orthopedic surgery
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to determine the safety of epoetin alfa and to determine the effectiveness of epoetin alfa in reducing the need for blood transfusions after major orthopedic surgery. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Patients undergoing major orthopedic surgery frequently require blood transfusions both during and after the operation. Agents that can increase the rate of red blood cell production would reduce the need for blood transfusions. Epoetin alfa is a genetically engineered form of a natural hormone, erythropoietin, that stimulates red blood cell production. This is a randomized, double-blind, placebo-controlled, parallel group, multicenter study. The study compares the effectiveness of epoetin alfa in reducing the need for blood transfusions in patients who are expected to require at least 2 units of blood following major orthopedic surgery. Eligible patients will be randomly assigned to receive either epoetin alfa (100 or 300 U/kg, depending upon their body weight) or a matching placebo, by injection beneath the skin starting 10 days before scheduled surgery, on the day of surgery (after surgery), and for 4 days after surgery. Additionally, all patients will start taking an oral iron supplement at least 10 days before their scheduled surgery. Effectiveness will be determined by the number of transfusions required following surgery, and on changes in hematocrit (iron-containing pigment in red blood cells), hemoglobin (oxygen-carrying component of red blood cells), and reticulocyte (immature red blood cells) levels from the start of the study to the end of the study. Safety evaluations will include the incidence and severity of adverse events, and changes in clinical laboratory tests, vital signs, and physical examination findings throughout the study. The study hypothesis is that patients treated with epoetin alfa will require fewer blood transfusions after surgery than patients treated with placebo. Epoetin alfa (300 U/kg or 100 U/kg), or matching placebo, by injection beneath the skin beginning 10 days before scheduled surgery and ending 4 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for major orthopedic surgery who are expected to require transfusion of at least 2 units of red blood cells
* who are unwilling or unable to participate in a transfusion program wherein a patient's own blood is donated before surgery
* having no significantly abnormal blood or urine test results
* having a hematocrit <= 45%

Exclusion Criteria:

* Patients with any blood disease, significant heart and blood vessel disease or signs and symptoms of other significant disease and/or dysfunction
* having signs and symptoms of significant and ongoing blood loss
* having a seizure disorder, uncontrolled high blood pressure, or infections or cancers that may make it difficult to respond to the study drug
* received medication known to suppress the formation of red blood cells within 1 month before the start of the study
* received a blood transfusion within 1 month before the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 1991-04; Study Completion 1991-10 (Actual)

PRIMARY OUTCOMES:
Transfusion requirements following surgery; Changes in hematocrit, hemoglobin, and reticulocyte count from the start of the study to the end of the study

SECONDARY OUTCOMES:
Adverse events; Changes in clinical laboratory test results, vital signs, and physical examination findings

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study to determine the safety of epoetin and whether epoetin alfa can reduce the need for blood transfusion in patients after major orthopedic surgery — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=680&filename=CR005902_CSR.pdf